CLINICAL TRIAL: NCT06213350
Title: Athlete Needs Assessment & Focus Groups
Status: Recruiting | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Tiffany Stewart, Professor, Pennington Biomedical Research Center
Other Study IDs: PBRC 2023-075
Record Dates: First submitted 2023-12-19; First posted 2024-01-19 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Athlete Support

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Needs Assessment Participants
- Focus Group Participants

SUMMARY:
The overall objective of this study is to investigate various physical and mental health needs of collegiate athletes and how they differ in and out of sport. Researchers aim to identify facets of support that athletes may need when transitioning out of sport. To achieve this objective, the study is broken down into two specific parts: 1) an online, anonymous survey assessing 200 athletes to evaluate support needed both during and post sport, quantitatively; and 2) focus groups with 50 athletes who are about to retire or have retired from sport recently to evaluate support needed both during and post sport, qualitatively.

ELIGIBILITY:
Inclusion Criteria:

* Current and previous collegiate athletes over the age of 18 and within two years before leaving sport or within five years after leaving sport.

Exclusion Criteria:

* Athletes under the age of 18 and not within two years before or five years after leaving sport will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Current and previous collegiate athletes over the age of 18 and within two years before leaving sport or within five years after leaving sport.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-02-27 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Qualitative Feedback | 1 year
  Responses to guided open ended questions

CONTACTS AND LOCATIONS:
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No